CLINICAL TRIAL: NCT01525745
Title: Randomized Ph II Study of Stereotactic Body Radiotherapy (SBRT) Versus Conventional Radiation for Spine Metastasis
Brief Title: Randomized Study of Stereotactic Body Radiotherapy vs. Conventional Radiation for Spine Metastasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Local IRB decision due to poor accrual
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Anand Mahadevan, Principle Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-294
Record Dates: First submitted 2011-12-13; First posted 2012-02-03 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Primary Tumor; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiosurgery/SBRT (Active Comparator): Radiosurgery/SBRT
  Interventions: Radiation: Radiosurgery/SBRT
- External Beam Radiation Therapy (Active Comparator): External Beam Radiation Therapy
  Interventions: Radiation: External Beam Radiation Therapy

INTERVENTIONS:
Radiation: Radiosurgery/SBRT — 1, 3 or 5 SBRT treatments
  Arms: Radiosurgery/SBRT
Radiation: External Beam Radiation Therapy — 10 consecutive days of standard radiation
  Arms: External Beam Radiation Therapy

SUMMARY:
The purpose of this study is to determine how effective SBRT is compared to traditional radiation in treating the cancer that has spread to your spine and is causing pain. SBRT is delivered at a higher dose for a shorter period of time when compared to standard radiation therapy and the aim is to see if there will be an improvement both in pain control and your cancer It is not known whether SBRT is better or worse than current standard therapy. If you are selected to receive the experimental treatment in this research study, SBRT uses highly focused x-rays that deliver a single high dose to a specific area of the spine compared to conventional standard radiation over a period of 10 days which has been the standard proven treatment to help your condition. The investigators will also determine which treatment provides the most rapid pain relief with the least side effects. It is possible that SBRT may not be better or could be more toxic. The investigators will conduct quality of life assessments and pain scale index to assess how you are feeling once you have had the intervention.

DETAILED DESCRIPTION:
Randomization means that you are put into a group by chance. It is like flipping a coin. Neither you nor the research doctor will choose what group you will be in.

You will have a 2 to 1 chance of being placed in the SBRT to standard radiation group. Since SBRT is the newer treatment being tested, we would like to include more patients in this group.

Treatment Procedures:

SBRT: You may receive one, three or five SBRT treatments depending on the extent of your cancer. During each treatment you will be assessed by a nurse and a physician for a physical and neurological assessment. The treatment itself would last approximately I hour where you will be lying on a treatment table. Prior to each treatment you will have a physical and neurological assessment by a physician. Standard Radiation: You will receive ten consecutive working days of standard radiation. While each treatment lasts five to ten minutes, the entire visit may last up to thirty minutes. During the treatment you will be lying on a treatment table. Once per week you will have a physical and neurological assessment by your treating physician After the final treatment of the study therapy: We would like to keep track of your medical condition for at least 12 months after you receive treatment. We would like to do this by having you come in to the clinic at months 1, 3, 6, 12 and 24 months after treatment*. At these visits we will be looking for the same information as during the screening time frame. This includes:

* A history and physical from you
* A Performance Status of how you are able to carry on with your usual activities.
* A Pain scale questionnaire called the Numerical Rating Pain Scale(NRPS) that asks to explain your pain symptoms on a 0-10 scale
* 3 Quality Of Life (QOL) Assessments described below:
* Functional Assessment of Cancer Therapy-General (FACT-G)
* The Brief Pain Inventory (BPI)
* The EuroQOL (EQ-5D)
* An assessment of your tumor by MRI (Magnetic Resonance Imaging)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary tumor or metastatic cancer with radiological diagnosis of spine metastasis
* The patient must have localized spine metastasis from the C1 to L5 levels by a screening imaging study
* Zubrod Performance Status 0-2
* History/physical examination within 2 weeks prior to registration
* Negative pregnancy test within 2 weeks prior to registration for women of childbearing potential
* Women of childbearing potential and male participants who are sexually active must agree to use a medically effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* MRI of the involved spine within 4 weeks prior to registration to determine the extent of the spine involvement
* Numerical Rating Pain Scale within 1 week prior to registration; the patient must have a score on the Scale of >5 for at least one of the planned sites for spine radiosurgery. Patients taking medication for pain at the time of registration are eligible.
* Neurological examination within 1 week prior to registration to rule out rapid neurologic decline

Exclusion Criteria:

* Histology of myeloma, lymphoma or germ cell tumors.
* Non-ambulatory patients
* Spine instability due to a compression fracture
* > 50% loss of vertebral body height
* Frank spinal cord displacement or epidural involvement with> 25% encirclement of cord or >25% spinal canal involvement.
* Prior radiation to the index spine
* Patients for whom an MRI of the spine is medically contraindicated
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Mahadevan, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Beth Israel Deacness Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all participants were enrolled in the RadOnc clinic at BIDMC
Period: Overall Study
Arm/Group | Radiosurgery/SBRT | External Beam Radiation Therapy
Started | 4 | 2
Completed | 3 | 1
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- A/Radiosurgery-SBRT: Radiosurgery/SBRT: 1, 3 or 5 SBRT treatments
- B/External Beam Radiation Therapy: External Beam Radiation Therapy: 10 consecutive days of standard radiation
- Total: Total of all reporting groups
Arm/Group | A/Radiosurgery-SBRT | B/External Beam Radiation Therapy | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pain Control as Measured by NPRS
Description: Determine if image-guided radiosurgery/SBRT improves pain control as measured by NPRS as compared to conventional external beam radiotherapy
Time Frame: 2 years
Population: study was terminated by the local IRB due to slow accrual. 1 participant withdrew consent and 1 participant did not complete the assigned arm treatment per protocol and then removed from study. left with 4 participants and data were not collected for any participants therefore no analysis has been done.
Arm/Group | A/Radiosurgery-SBRT | B/External Beam Radiation Therapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Duration of Pain Response
Description: Determine if image-guided radiosurgery/SBRT improves duration of pain as compared to conventional external beam radiotherapy
Time Frame: 2 years
Population: data not collected, therefore no analysis done
Arm/Group | Radiosurgery/SBRT | External Beam Radiation Therapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life
Description: Evaluate potential benefit of image-guided radiosurgery/SBRT on change in and overall quality of life as measured by FACT-G, BPI and EQ-5D
Time Frame: 2 years
Population: data not collected, therefore no analysis done
Arm/Group | A/Radiosurgery-SBRT | B/External Beam Radiation Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Long Term Effects of Image-guided Radiosurgery/SBRT
Description: Long term effects of image-guided radiosurgery/SBRT on the vertevral bone and spinal cord
Time Frame: 2 years
Population: data not collected, therefore no analysis done
Arm/Group | A/Radiosurgery-SBRT | B/External Beam Radiation Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Survival
Description: Progrsesion Free and Overall Survival
Time Frame: 2 years
Population: data not collected, therefore no analysis done
Arm/Group | A/Radiosurgery-SBRT | B/External Beam Radiation Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were monitored but none occurred.
Arm/Group | A/Radiosurgery-SBRT | B/External Beam Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No